CLINICAL TRIAL: NCT00966290
Title: Anticoagulant Clinic-based Shared-care Versus Usual Cate Management of Vitamin K Antagonist Therapy : the Open, Randomized Multicenter Study
Brief Title: Anticoagulant Clinics and Vitamin K Antagonists
Acronym: COMPARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: LLAU ME, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0200301; PHRC 2002
Record Dates: First submitted 2009-08-21; First posted 2009-08-26 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Blood Coagulation Disorders
Keywords: anticoagulants; management; anticoagulation clinics; randomized comparison
MeSH Terms: conditions — Blood Coagulation Disorders | interventions — Anticoagulants; Warfarin; Acenocoumarol; fluindione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACC group (Experimental): Anticoagulant clinic-based shared-care group
  Interventions: Drug: Anticoagulant (warfarin, acenocoumarol, fluindione)
- UC group (Active Comparator): Usual care group
  Interventions: Drug: Anticoagulant (warfarin, acenocoumarol, fluindione)

INTERVENTIONS:
Drug: Anticoagulant (warfarin, acenocoumarol, fluindione) — Anticoagulant clinic based shared-care group
  Other Names: Patients whose anticoagulation is managed by the general practitioner in collaboration with anticoagulant clinic
  Arms: ACC group
Drug: Anticoagulant (warfarin, acenocoumarol, fluindione) — Usual care group
  Other Names: Patients whose anticoagulation is managed by the general practitioner
  Arms: UC group

SUMMARY:
Background: Whether the management of vitamin K antagonists (VKA) therapy by general practitioners with the collaboration of anticoagulation clinics (ACC) provides better clinical outcomes than that accomplished by general practitioners alone (usual care [UC] management) is not clear.

Objectives: To compare ACC-based shared-care management with UC management of VKA therapy with respect to clinical events.

Patients/Methods: Open, randomized, multicenter study in patients starting VKA therapy for at least three months. The primary study outcome is a composite of confirmed symptomatic thromboembolic or major bleeding events. All-cause mortality is a secondary outcome. All outcomes are reviewed by a central, independent adjudication committee.

DETAILED DESCRIPTION:
Study design

The COMPARE (Comparison of Oral anticoagulation Monitoring Practice: A Randomized Evaluation) study is an open, centrally randomized, multicenter, prospective, controlled study comparing two models of vitamin K antagonist (VKA) therapy management. Written informed consent is obtained from each patient and general practitioner before randomization.

Setting and participants

The study concerned patients referred to the anticoagulation clinic (ACC) of various University Hospitals in France. Eligible patients are consecutive patients who were starting a course of VKA therapy scheduled to last for at least three months.

Randomization and interventions

All eligible patients are evaluated by a physician specialized in vascular medicine or hematology. After their demographic characteristics and medical history had been recorded, they are randomized to one of the models of VKA therapy management, either UC management or ACC-based shared-care management. Randomization is stratified by center; the list of randomization is computer-generated according to a permuted block design with a block size of four, six or eight. General practitioners are informed of the outcome of randomization by a standardized letter. In patients randomized to the UC management group, the monitoring of VKA therapy is left to the general practitioner's discretion according to his/her preferences and habits. Patients randomized to the ACC-based shared-care management group receive a standardized educational package; moreover, each biological laboratory measuring INR values for the patients of this group is contacted to explain the importance of rapid restitution of the results. A computer-generated dose proposal is also given, both by telephone and by fax, to the general practitioners who follow up patients randomized to the ACC-based shared-care management group; however, they were free to accept or ignore this proposal. All patients receive a logbook in which to record their INR results.

Study outcomes

The primary study outcome is a composite of symptomatic and objectively confirmed thromboembolic or major bleeding events at 18 months. Thromboembolic events are acute myocardial infarction, stroke, peripheral arterial occlusion, deep-vein thrombosis or pulmonary embolism. Major bleeding events are fatal bleeding, or any bleeding leading to functional impairment or requiring hospitalization. All-cause mortality is a secondary outcome measure. All outcomes are reviewed by a central, independent adjudication committee, the members of which were unaware of the patients' study group.

The quality of anticoagulation control is evaluated in all randomized patients with at least two INR measurements. This parameter is assessed by determining (1) the percentage of INR within the target range, (2) the percentage of time during which the INR was within the target range in relation to the total length of the observation period, according to the linear interpolation method, and (3) the variability index (σ2).

Statistical analysis

This is a superiority study in which we hypothesize that ACC-based shared-care management would reduce the cumulative incidence of the primary study outcome by 50% compared with UC management. On the basis of previous non-controlled studies, we assumed that the cumulative incidence of the primary study outcome would be 10% in patients assigned to the UC management group. Given these assumptions, we calculated that the recruitment of 600 patients per group would allow confirmation of the statistical hypothesis with 90% power and a two-sided, type I error of 0.05.

The statistical analyses will be performed on all randomized patients on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* inpatients and outpatients who are starting a course of VKA therapy scheduled to last for at least three months

Exclusion Criteria:

* life expectancy of less than three months
* contraindication to anticoagulant therapy because of bleeding risk
* refusal of his/her general practitioner to participate in the study
* no general practitioner likelihood of poor follow-up or poor compliance (e.g., patients unable to care for themselves, lacking adequate home support or unwilling to comply with the treatment care plan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1006 (Actual)
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Each patient is contacted by standardized telephone calls every three months to determine whether he/she has experienced any thromboembolic or major bleeding complication, and to identify any interruptions in VKA treatment | Patients are followed up for the duration of VKA treatment until 12 months or plus three days after treatment discontinuation

SECONDARY OUTCOMES:
Quality of anticoagulation control evaluated in all patients with at least two INR measurements and assessed by determining (1) the percentage of INR within the target range, (2) the percentage of time during which the INR is within the target range | Patients are followed up for the duration of VKA treatment until 12 months or plus three days after treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Henri Boccalon, MD, Principal Investigator — University Hospital, Toulouse; Alessandra BURA-RIVIERE, MD, Study Director — University Hospital, Toulouse; Patrick Mismetti, MD, Study Director — University Hospital Saint-Etienne; Bernard Boneu, MD, Study Director — University Hospital, Toulouse
Locations (7):
- France (7):
  - University Hospital, Brest
  - Louis Pasteur Hospital, Dole
  - University Hospital, Lille
  - Dupuytren University Hospital, Limoges
  - Bellevue University Hospital, Saint-Etienne
  - University Hospital, Strasbourg
  - Rangueil University Hospital, Toulouse